CLINICAL TRIAL: NCT00397280
Title: Innate Immunity Signal Transduction in Human Leukocytes
Brief Title: Immune Cell Response to Stimuli
Status: Recruiting | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070023; 07-E-0023
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-05-02

CONDITIONS: Inflammation
Keywords: Inflammatory Response; Lipopolysaccharide; Natural History
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Any healthy donors meeting inclusion/exclusion criteria

SUMMARY:
This study will investigate the response of immune cells (neutrophils, monocytes) to various signals in the test tube to determine how they sense the signals in the body and what substances they produce in response to them. It will determine how the cells may, under certain circumstances, contribute to inflammation, and will measure substances in the blood plasma (the liquid, non-cellular part of the blood) that might stimulate white blood cells, in order to understand how the blood responds to possible disease-related conditions.

Healthy normal volunteers 18 years of age and older who weigh at least 110 pounds may be eligible for this study. Participants give about 320 milliliters (mL) of blood (about 1 1/3 cups) or less at each donation. They donate no more than once every 8 weeks and no more than six times a year. On some occasions, less than 320 mL of blood may be drawn. The collected blood is separated into its components and specific cells are exposed to substances to examine their response.

DETAILED DESCRIPTION:
The objective of this study is several-fold. We wish to determine the response of white blood cells (neutrophils, monocytes, eosinophils, lymphocytes) to various signals in the test tube, to test how they sense the signals in the body, and what substances they produce. We wish to determine how these cells may, under certain circumstances, contribute to inflammation. We wish to measure the substances in the blood plasma that might contribute to stimulation of white blood cells to understand the response of the whole blood to potential disease-associated conditions.

The objective is to define the signaling pathways activated by lipopolysaccharide (LPS) and other selected innate immunity stimuli, and the downstream inflammatory functional consequences, in human leukocytes in vitro. Adult (18-65 yrs. old), nonpregnant, healthy volunteers will have 320 ml of whole blood collected by venipuncture in a monitored setting no more frequently than once every 8 weeks. No further interventions will be exercised upon the subjects. The whole blood will be fractionated into neutrophil, red blood cell, mononuclear cell, and plasma fractions using plasma-Percoll discontinuous centrifugation. Leukocytes will be subjected in vitro to inflammatory stimuli (e.g., LPS), and selected signaling outcomes (e.g., mitogen-activated protein kinase activation, Rho GTPase activation, protein-protein interactions) and functional measures (e.g., chemotaxis, superoxide anion and cytokine production) quantified in the absence and presence of relevant chemical inhibitors (e.g., SB203580, a p38 MAPK inhibitor). In each such experiment, cells from the daily donor will be used as paired controls to the in vitro experimental intervention (e.g., SB203580 inhibitor vs. DMSO vehicle). Three or more repetitions (on different donors) of each specific experimental outcome, as necessary, will be performed to establish statistical significance of findings.

A specific focus of the studies planned will be to define the role of lipid raft membrane microdomains in transduction of the LPS signal in human leukocytes. Lipid rafts are cholesterol-rich microdomains in the plasma membrane, within which the LPS receptor, Toll-like Receptor 4 (TLR4), has been described to reside. LPS signaling has been reported to be sensitive to raft cholesterol content, presumably because the specific repertoire of proteins in rafts is sensitive to raft cholesterol content. Rafts are thought to act as dynamic signaling platforms for co-segregation of proximal adaptor proteins, kinases, and other signaling proteins. Of interest, while LPS has been described to modulate the activity of proteins that determine raft cholesterol content (egg, Liver X Receptor, ABCA1), virtually no work has been done to clarify: 1) the mechanisms underlying LPS-induced intracellular cholesterol redistribution, and, more importantly, 2) whether such intracellular redistribution of cholesterol is causal to the signaling events triggered by LPS, or 3) whether innate immunity signaling is dependent upon inter-subject variations in raft cholesterol content.

Furthermore, we will investigate the role of the tumor suppressor gene p53 in the regulation of inflammation. It is now widely accepted that inflammation and cancer development are interconnected. Dr. Menendez is one of the international leaders in the study of the tumor suppressor gene p53. His group has discovered that activation of p53 through exposure to carcinogenic stimuli leads to differential expression of genes that have a direct effect on the inflammatory response, such as several toll-like-receptor genes. Dr. Menendez will use human leukocytes that will be isolated from whole blood. He will expose these cells to stimuli that activate p53, such as doxorubicin (a chemotherapy agent) or radiation, and examine the expression of toll-like-receptor genes as well as the response to LPS and other inflammatory agents in vitro.

Finally, we will investigate the role of zinc-finger proteins in gene expression in inflammatory cells. ZFP36 is an RNA binding zinc finger protein that is involved in the turnover of mRNAs encoding several clinical important cytokines, including TNFa. Several missense, promoter and 3'-untranslated variants have been identified in humans; in some cases, these variants and their haplotypes have been associated with human inflammatory disease. We will isolate peripheral blood macrophages and stimulate them with LPS and other cytokines, then evaluate the behavior of cytokine mRNA and gene expression.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Normal, healthy adult donors as judged by screening questionnaire
* Nonpregnant
* Weighing at least 110 lbs
* 18-65 years of age
* HIV negative (proof required every 6 months we will conduct test)*
* Hepatitis B surface antigen and hepatitis C serology negative (checked every 6 months we will conduct test)*

  * The rationale for HIV and hepatitis viral testing is that chronic viral infection may alter and possibly invalidate our experimental results. HIV and hepatitis results will be confidentially obtained. Testing will be contracted to an external certified laboratory and will be paid for by the study group. Results will be available only to the study doctor/PI (Fessler), the study coordinator, the CRU Director (Garantziotis, LAI), and the donor, with the few caveats that follow

All positive HIV, hepatitis B, and hepatitis C results will be promptly communicated to the donor by the study doctor/PI or the CRU Director. The participant will be referred to their physician and/or to the N.C. Department of Health for confirmatory testing and counseling. As explained in detail in the attached Supplement describing N.C. State Department of Health code will be followed. The state code mandates reporting of positive results along with the participant s name and identifying information to the N.C. Department of Public Health. Upon contracting with the testing laboratory, clarification will be obtained and documented as to whether the contracted laboratory or the study MD will be responsible for reporting positive results to the state to avoid duplication of reporting. Upon receipt of the test results, the N.C. Department of Health will contact the participant to inform them of the positive result, how to find care, how to avoid infecting others, how the newly diagnosed HIV and/or hepatitis infection is reported, and the importance of informing their partners at possible risk because of their HIV and/or hepatitis infection. If the HIV, hepatitis B, and hepatitis C results are negative, the participant will be not be notified. However, the participant may contact the research study nurse for their results.

HIV and hepatitis B/C test results, non-reactive and reactive, will be documented confidentially by the PI or study coordinator in the subject s file, and kept in a locked file cabinet in the CRU Medical Records Room.In order to document the reporting procedure and the time associated with the reporting process, a document has been created and placed in the study specific manual (Hepatitis B/C and HIV Notification Process for Reactive Results Form)

EXCLUSION CRITERIA:

By questionnaire:

Feeling ill within the last 24 hours.

Alcohol consumption in the last 24 hours.

Visit to the dentist in the last 24 hours.

A doctor visit for illness or vaccination in the last 2 weeks.

Diarrhea in the last 2 weeks.

Recurrent fever (4 weeks).

Pregnant or suspected pregnancy in the last 6 weeks.

Blood or plasma donation that will cause the participant to exceed 550ml of blood in the last 8 weeks.

Receiving a blood donation in the past 12 months.

Bleeding disorder.

Anemia.

Heart problems.

Insulin dependent diabetes.

Problems with blood donation.

Risk of or evidence of Creutzfeldt-Jacob Disease in the family.

HIV-positive status, Hepatitis B/C-positive status or other confirmed or suspected immunosuppressive or immunodeficient conditions.

Use of immunosuppressants or other immune-modifying drugs.

Use of selected medications within the preceding 5 days unless the PI or AI receiving the samples states otherwise (NSAIDS/aspirin/tylenol, antidepressants, antihistamines , corticosteroids, HMG CoA reductase inhibitors, and antihypertensives).

By exam:

Temperature over 99.5 F.

Blood pressure less than 90/50.

Blood pressure higher than 170/95 mm Hg.

Pulse rate less than 50 or greater than 100 beats/minute.

If blood donation exceeds 200ml:

* Hematocrit less than 34% for women or less than 36% for men, or greater than 56% for either gender.
* Patients will be informed of disqualifying vital signs and hematocrit values and advised by trained staff, as appropriate, to seek assistance from their physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any healthy donors meeting inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2009-07-13 (Actual)

PRIMARY OUTCOMES:
The objective is to define the signaling pathways activated by lipopolysaccharide (LPS) and other selected innate immunity stimuli, and the downstream inflammatory functional consequences, in human leukocytes in vitro. | analysis of the study
  The objective is to define the signaling pathways activated by lipopolysaccharide (LPS) and other selected innate immunity stimuli, and the downstream inflammatory functional consequences, in human leukocytes in vitro.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Fessler, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
It isn t known yet if there will be a plan to make IPD available

REFERENCES:
- [Background] Walker TS, Tomlin KL, Worthen GS, Poch KR, Lieber JG, Saavedra MT, Fessler MB, Malcolm KC, Vasil ML, Nick JA. Enhanced Pseudomonas aeruginosa biofilm development mediated by human neutrophils. Infect Immun. 2005 Jun;73(6):3693-701. doi: 10.1128/IAI.73.6.3693-3701.2005. PMID 15908399
- [Background] Fessler MB, Arndt PG, Frasch SC, Lieber JG, Johnson CA, Murphy RC, Nick JA, Bratton DL, Malcolm KC, Worthen GS. Lipid rafts regulate lipopolysaccharide-induced activation of Cdc42 and inflammatory functions of the human neutrophil. J Biol Chem. 2004 Sep 17;279(38):39989-98. doi: 10.1074/jbc.M401080200. Epub 2004 Jul 15. PMID 15262974
- [Background] Frasch SC, Henson PM, Nagaosa K, Fessler MB, Borregaard N, Bratton DL. Phospholipid flip-flop and phospholipid scramblase 1 (PLSCR1) co-localize to uropod rafts in formylated Met-Leu-Phe-stimulated neutrophils. J Biol Chem. 2004 Apr 23;279(17):17625-33. doi: 10.1074/jbc.M313414200. Epub 2004 Feb 6. PMID 14766753
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2007-E-0023.html